CLINICAL TRIAL: NCT02460991
Title: A Randomized Controlled Trial of Transcatheter Arterial Chemoembolization With Drug Eluting Beads (DEB-TACE) Versus Sorafenib in the Treatment of Unresectable, Locally Advanced Hepatocellular Carcinoma
Brief Title: A Study of ONCO-DOX in Locally Advanced Hepatocellular Carcinoma
Acronym: SOLACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLACE
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB-TACE (Experimental): ONCO-DOX (Doxorubicin loaded Microspheres) up to 150 mg per treatment; treatments can be repeated every 4-8 weeks until complete tumor response is achieved.
  Interventions: Device: DEB-TACE
- Sorafenib (Active Comparator): 200 mg Sorafenib twice daily; continue until unacceptable toxicity or unequivocal tumor progression
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Device: DEB-TACE
  Other Names: ONCO-DOX
  Arms: DEB-TACE
Drug: Sorafenib
  Other Names: Nexavar
  Arms: Sorafenib

SUMMARY:
This is a prospective, multicenter study that will be conducted at up to 40 centers in the United States and Outside United States (OUS). Participants in the study will be randomly assigned to receive either ONCO-DOX or sorafenib treatment. This study will evaluate the study participants' outcomes (medical condition) after being treated with ONCO-DOX and compare it to those treated with sorafenib alone.

DETAILED DESCRIPTION:
This is a prospective, two-arm, stratified then randomized (1:1), open label, controlled, multicenter Phase III trial to evaluate the safety and efficacy of ONCOZENE™ Microspheres loaded with doxorubicin (ONCO-DOX) in comparison with orally administered sorafenib in patients with unresectable, locally-advanced hepatocellular carcinoma (HCC).

Patients will be stratified by ECOG Performance Status 0 versus 1, portal vein invasion (yes vs. no), and alpha feto protein <400 versus ≥400. They will then be randomized at each site within each stratum.

The study will be conducted at up to 40 centers in the United States, Europe & Asia. Enrolled patients will be randomized with equal allocation by study site.

Patients will be followed for two years after the onset of treatment.

The study will assess prospectively the efficacy and safety of DEB-TACE (ONCO-DOX) in patients with unresectable, locally-advanced HCC. The primary objective of this study is to compare the overall survival between DEB-TACE (ONCO-DOX) and sorafenib treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. ≥18 years of age
3. Diagnosis of HCC
4. Locally advanced HCC
5. Preserved liver function
6. Eastern Cooperative Oncology Group 0 or 1

Exclusion Criteria:

1. Presence of extra-hepatic spread of disease.
2. Macrovascular invasion of lobar portal vein branches or main portal vein.
3. Candidate for surgical resection, transplantation, or local ablation.
4. Prior intra-arterial embolization, chemotherapy or systemic therapy for HCC.
5. Any contraindication for TACE.
6. Platelet count <50,000/mm3 or international normalized ratio >1.5.
7. Previous treatment with anthracycline antibiotics (e.g. Doxorubicin) or sorafenib.
8. Unstable coronary artery disease or recent myocardial infarct (i.e. within 1 year).
9. Known ejection fraction < 50%.
10. Current infections requiring antibiotic therapy.
11. Suffering from a known bleeding disorder.
12. Renal insufficiency (serum creatinine > 2 mg/dL).
13. Aspartate aminotransferase and/or alanine transaminase >5 times upper limit of normal.
14. Presence of advanced liver disease.
15. Any contraindication for doxorubicin administration:
16. Any co-morbid condition or social situation, which has a high likelihood of causing poor compliance with the study protocol or jeopardizes the patient's safety.
17. Patient has another primary tumor, with the exception of conventional basal cell carcinoma, superficial bladder cancer, melanoma in situ, or treated prostate cancer currently without biochemical or radiographic evidence of active disease
18. Participation in a clinical trial of an investigational device or drug within 4 weeks of study entry.
19. Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Becker, Study Director — Boston Scientific Corporation
Locations (6):
- United States (6):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- DEB-TACE: ONCO-DOX (Doxorubicin loaded Microspheres) up to 150 mg per treatment; treatments could be repeated every 4-8 weeks until complete tumor response was achieved.
- Sorafenib: 200 mg of Sorafenib twice daily; continue until unacceptable toxicity or unequivocal tumor progression
Period: Overall Study
Arm/Group | DEB-TACE | Sorafenib
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only two subjects were randomized prior to the suspension of the study. Both subjects were randomized to the Sorafenib arm of the study. No subjects were randomized to DEB-TACE.
Groups:
- Total: Total of all reporting groups
Arm/Group | DEB-TACE | Sorafenib | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2
Age [Mean (Full Range); unit: years] |  | 63 [56 to 70] | 63 [56 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival in HCC subjects with minimum follow-up of subjects to at least one year
Time Frame: 1 year
Population: The planned analyses were not performed due to early termination.
Arm/Group | DEB-TACE | Sorafenib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) determined by radiological assessment using mRECIST criteria
Time Frame: 2 years
Population: The planned analyses were not performed due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | DEB-TACE | Sorafenib
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

3. Secondary Outcome: Time to Extrahepatic Spread
Description: Time to Extrahepatic Spread for each subject
Time Frame: 2 years
Population: The planned analyses were not performed due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | DEB-TACE | Sorafenib
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

4. Secondary Outcome: Proportion Progression Free
Description: Proportion Progression-Free (PPF) at one year
Time Frame: 1 year
Population: The planned analyses were not performed due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | DEB-TACE | Sorafenib
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

5. Secondary Outcome: Frequency of Treatment Emergent Adverse Events
Description: The frequency of treatment emergent adverse events at 30 day, 3, 6, 9, 12, 18, and 24-months following the initial treatment. The proportions of patients in each arm experiencing treatment emergent adverse events will be presented descriptively with the number experiencing the event, the number evaluated, the percentage, and the exact two-sided 95% confidence interval.
Time Frame: 2 years
Population: Study was terminated early. Adverse events were captured through the end of the study.
Measure: Number; unit: participants
Groups:
- DEB-TACE: ONCO-DOX (Doxorubicin loaded Microspheres) up to 150 mg per treatment; treatments can be repeated every 4-8 weeks until complete tumor response is achieved.
  DEB-TACE
- Sorafenib: 200 mg Sorafenib twice daily; continue until unacceptable toxicity or unequivocal tumor progression
  Sorafenib
Arm/Group | DEB-TACE | Sorafenib
Number analyzed (Participants) | 0 | 2
participants |  | 2

6. Other Pre Specified Outcome: Proportion Achieved Tumor Response
Description: The proportion of patients in each group that achieve complete response (CR), partial response (PR), and stable disease (SD) will be presented and compared across treatment groups.
Time Frame: 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: FACT-Hep Quality of Life
Description: FACT-Hep quality of life instrument validated in patients with Hepatic cancer.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Description: Only two subjects were randomized prior to the suspension of the study and both were randomized to the Sorafenib arm. No subjects were randomized to DEB-TACE.
Arm/Group | DEB-TACE | Sorafenib
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2
Other Adverse Events (participants affected / at risk) | 0/0 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEB-TACE (N=0) | Sorafenib (N=2)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEB-TACE (N=0) | Sorafenib (N=2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Desquamation of bottom of feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Internal Hemorroids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight Loss (Investigations) | 0 (0) | 1 (1)
Lung Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The planned analyses were not performed due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02460991/Prot_SAP_ICF_000.pdf